CLINICAL TRIAL: NCT03569020
Title: Dietary Approaches to Stop Hypertension (DASH) Diet Effects on Serum Uric Acid (SUA) in Adults With Hyperuricemia and Gout
Brief Title: The Diet Gout Trial
Acronym: DIGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Harvard Medical School (HMS and HSDM) (Other); Rheumatology Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00153409
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2019-11

CONDITIONS: Gout; Hyperuricemia
Keywords: Diet; Nutrition; DASH; Gout; Hyperuricemia; Potassium; Uric acid; Trial; Blood pressure; Glucose; Lipid; Cholesterol; Weight; Arthritis; BMI; Body mass index; Fruit; Vegetable; Low fat dairy; Lean meat; Fiber
MeSH Terms: conditions — Gout; Hyperuricemia; Body Weight; Arthritis

STUDY DESIGN:
Intervention Model Description: Half of participants will be randomly assigned 1 of 2 potential sequences. All participants will ultimately participate in each study period, but the order will be randomly assigned 1:1.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators will not know which assignment the participants were given. The laboratory measuring uric acid will not know which intervention the participants were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietitian-Directed Diet (Experimental): Participants will be provided $105/week ($15/day) to purchase foods in servings that correspond to the DASH diet and thus include fruits, vegetables, lean meat, low fat dairy, and high fiber foods. Participants will also be asked to restrict red meat, sweets, and sugary beverages during this intervention period. A dietitian will help participants order foods from a digital supermarket. Foods will be delivered to the Johns Hopkins ProHealth Research Clinic for weekly pick-up. This study period will last 4 weeks.
  Interventions: Other: Subsidy for food purchases and dietitian education
- Self-Directed Diet (No Intervention): Participants will be asked to consume their typical diet for 4 weeks. There will be no subsidy during this period.

INTERVENTIONS:
Other: Subsidy for food purchases and dietitian education — $105/wk of DASH-like foods over 4 weeks purchased with the help of a dietitian in a proportion that reflects the DASH diet.
  Arms: Dietitian-Directed Diet

SUMMARY:
Unhealthy diet has long been associated with high uric acid levels and gout. The DASH diet may lower uric acid levels. This study will examine the effects of the DASH diet on uric acid in adults with a history of gout.

DETAILED DESCRIPTION:
The public health burden of gout is substantial. Several lines of evidence suggest that a DASH diet might lower uric acid. However, there are no trials of the DASH diet in adults with gout. This trial is a cross-over study of the effects of a DASH-like diet on uric acid in adults with gout and hyperuricemia, who are not taking urate-lowering therapy.

Perpetuated by the "Western" lifestyle and resulting obesity epidemic, the prevalence of gout has increased over the past few decades to 3.9% of US adults (8.3 million individuals). This prevalence increases with age to 9.3% of US adults over 60 years (4.7 million).

Participants will be community-dwelling adults, aged 18+ with a baseline serum uric acid level of 7 mg/dL, who have a self-reported history of gout and are not taking urate lowering medications (e.g. allopurinol, febuxostat, probenecid).

This trial is comprised of two study periods: (1) a dietitian-directed diet (DD) or (2) self-directed usual diet (SD). Each period lasts 4 weeks. All participants will participate in both periods, but half will undergo the dietitian-directed diet first while the other half will undergo the self-directed diet first. During the dietitian-directed diet, participants will receive $105/week of foods in a pattern that conforms to the DASH diet. The DASH diet emphasizes fruit, vegetables, lean meat, low fat dairy, and high fiber, while restricting red meat, sweets, and sugary beverages. During the self-directed diet, participants will be asked to eat their typical diet outside of the study. Investigators anticipate 40 participants in this study.

The primary outcome is uric acid. Secondary outcomes of this study include: body mass index, systolic and diastolic blood pressure, fasting cholesterol, and fasting blood glucose. Both primary and secondary outcomes will be measured 3 times: (1) before the study begins (baseline), (2) after period 1 (at 4 weeks), and (3) after period 2 (at 8 weeks). Patient-reported outcomes, dietary compliance, and urine electrolytes will be assessed throughout the study as well.

The primary comparison will be serum uric acid concentrations measured after the 4-week dietitian-directed diet versus uric acid concentrations measured after the 4-week self-directed diet (DD vs. SD). Comparisons will be made within person using generalized estimating equations (GEE) with and without adjustment for baseline uric acid concentration. Investigators will use GEE models for secondary outcomes as well.

ELIGIBILITY:
Inclusion Criteria:

Age > 18-100 years

Self-reported gout diagnosis

Serum Uric Acid > 7 mg/dL

Exclusion Criteria:

Recent or planned changes to urate lowering therapies (e.g. allopurinol, febuxostat, probenecid)

Recent or planned changes to hypertension, lipid, or diabetes medications

Patients with hyperkalemia (>5 mmol/L)

Chronic kidney disease (GFR < 30 cc/min), kidney transplant, dialysis

Gastro-intestinal conditions (e.g. history of gastric bypass surgery, active inflammatory bowel disease, malabsorption, or major GI resection)

Active cancer treatment (e.g. radiation or chemotherapy)

Diagnosis of any of the following in the past 6 months: heart attack, heart failure, angina, coronary bypass or angioplasty, or Chronic Obstructive Pulmonary Disease (COPD)

Alcohol use over 14 drinks per week

Inability to give informed consent

Active use of warfarin, insulin, or chronic steroids (like prednisone)

Terminal or mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 43 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Miller, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins ProHealth Research Clinic, Woodlawn, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghazi L, Drawz PE, Pajewski NM, Juraschek SP. The Association of Orthostatic Hypotension With Ambulatory Blood Pressure Phenotypes in SPRINT. Am J Hypertens. 2021 May 22;34(5):511-520. doi: 10.1093/ajh/hpaa184. PMID 33186448
- [Derived] Miller HN, Charleston J, Wu B, Gleason K, White K, Dennison Himmelfarb CR, Ford DE, Plante TB, Gelber AC, Appel LJ, Miller ER 3rd, Juraschek SP. Use of electronic recruitment methods in a clinical trial of adults with gout. Clin Trials. 2021 Feb;18(1):92-103. doi: 10.1177/1740774520956969. Epub 2020 Sep 15. PMID 32933342

RESULTS

PARTICIPANT FLOW:
Groups:
- Dietitian-Directed Diet Then Self-Directed Diet: During the dietitian-directed diet, participants will be provided $105/week ($15/day) to purchase foods in servings that correspond to the DASH diet and thus include fruits, vegetables, lean meat, low fat dairy, and high fiber foods. Participants will also be asked to restrict red meat, sweets, and sugary beverages during this intervention period. A dietitian will help participants order foods from a digital supermarket. Foods will be delivered to the Johns Hopkins ProHealth Research Clinic for weekly pick-up. This study period will last 4 weeks.
  Subsidy for food purchases and dietitian education: $105/wk of DASH-like foods over 4 weeks purchased with the help of a dietitian in a proportion that reflects the DASH diet.
  This is followed by 4-weeks of the self-directed diet (referent diet).
  During the self-directed diet, participants will be asked to consume their typical diet for 4 weeks. There will be no subsidy during this period. This is followed by the 4-week Dietitian-Directed Diet.
- Self-Directed Diet Then Dietitian-Directed Diet: During the self-directed diet, participants will be asked to consume their typical diet for 4 weeks. There will be no subsidy during this period. This is followed by the 4-week Dietitian-Directed Diet.
  During the Dietitian-Directed Diet, participants will be provided $105/week ($15/day) to purchase foods in servings that correspond to the DASH diet and thus include fruits, vegetables, lean meat, low fat dairy, and high fiber foods. Participants will also be asked to restrict red meat, sweets, and sugary beverages during this intervention period. A dietitian will help participants order foods from a digital supermarket. Foods will be delivered to the Johns Hopkins ProHealth Research Clinic for weekly pick-up. This study period will last 4 weeks.
  Subsidy for food purchases and dietitian education: $105/wk of DASH-like foods over 4 weeks purchased with the help of a dietitian in a proportion that reflects the DASH diet.
Period: Period 1
Arm/Group | Dietitian-Directed Diet Then Self-Directed Diet | Self-Directed Diet Then Dietitian-Directed Diet
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Dietitian-Directed Diet Then Self-Directed Diet | Self-Directed Diet Then Dietitian-Directed Diet
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a crossover design. Baseline characteristics are presented by participants' period 1 assignment.
Groups:
- Dietitian-Directed Diet Then Self-Directed Diet: Participants will be provided $105/week ($15/day) to purchase foods in servings that correspond to the DASH diet and thus include fruits, vegetables, lean meat, low fat dairy, and high fiber foods. Participants will also be asked to restrict red meat, sweets, and sugary beverages during this intervention period. A dietitian will help participants order foods from a digital supermarket. Foods will be delivered to the Johns Hopkins ProHealth Research Clinic for weekly pick-up. This study period will last 4 weeks.
  Subsidy for food purchases and dietitian education: $105/wk of DASH-like foods over 4 weeks purchased with the help of a dietitian in a proportion that reflects the DASH diet.
- Self-Directed Diet Then Dietitian-Directed Diet: Participants will be asked to consume their typical diet for 4 weeks. There will be no subsidy during this period.
- Total: Total of all reporting groups
Arm/Group | Dietitian-Directed Diet Then Self-Directed Diet | Self-Directed Diet Then Dietitian-Directed Diet | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: mg/dL] | 57.5 (13.3) | 60.5 (10.7) | 59.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 18 | 17 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 12 | 9 | 21
  White/Caucasian | 8 | 9 | 17
  Asian/Pacific Islander | 2 | 3 | 5
  Hispanic or Latino | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Uric Acid Level
Description: Measured in serum
Time Frame: Baseline
Population: This was a crossover design. All 43 participants underwent both interventions. The data is presented by first period assignment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dietitian-Directed Diet Then Self-Directed Diet | Self-Directed Diet Then Dietitian-Directed Diet
Number analyzed (Participants) | 22 | 21
mg/dL | 8.23 (0.74) | 8.03 (0.79)

2. Primary Outcome: Uric Acid Level
Description: Measured in serum
Time Frame: At 4-weeks
Population: This was a crossover study. Data are presented by first period assignment. The 4-week results represent period 1.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dietitian-Directed Diet | Self-Directed Diet
Number analyzed (Participants) | 22 | 21
mg/dL | 7.67 (1.25) | 8.03 (1.13)

3. Primary Outcome: Uric Acid Level
Description: Measured in serum
Time Frame: At 8-weeks
Population: This was a crossover design. Results are presented by period 1 assignment. The 8-week results represent the effect of the second period.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dietitian-Directed Diet | Self-Directed Diet
Number analyzed (Participants) | 22 | 21
mg/dL | 7.75 (1.15) | 7.98 (1.15)

4. Secondary Outcome: Systolic Blood Pressure (mm Hg)
Time Frame: Baseline, 4-weeks, 8-weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Dietitian-Directed Diet Then Self-Directed Diet | Self-Directed Diet Then Dietitian-Directed Diet
Number analyzed (Participants) | 22 | 21
mm Hg
  Baseline | 125.0 (17.0) | 123.5 (12.4)
  Period 1 (4-weeks) | 126.4 (15.2) | 123.7 (14.2)
  Period 2 (8-weeks) | 129.4 (17.2) | 124.8 (14.4)

5. Secondary Outcome: Diastolic Blood Pressure (mm Hg)
Time Frame: At baseline, 4-weeks, 8-weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Dietitian-Directed Diet Then Self-Directed Diet | Self-Directed Diet Then Dietitian-Directed Diet
Number analyzed (Participants) | 22 | 21
mm Hg
  Baseline | 74.9 (11.3) | 72.6 (10.5)
  Period 1 | 76.1 (11.9) | 75.0 (11.8)
  Period 2 | 77.3 (11.7) | 74.0 (11.4)

6. Secondary Outcome: Fasting Blood Glucose (mg/dL)
Description: Measured in serum
Time Frame: Baseline, 4-weeks, 8-weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dietitian-Directed Diet Then Self-Directed Diet | Self-Directed Diet Then Dietitian-Directed Diet
Number analyzed (Participants) | 22 | 21
mg/dL
  Baseline | 93.0 (11.6) | 103.0 (18.1)
  Period 1 | 96.5 (12.1) | 103.2 (27.7)
  Period 2 | 97.1 (12.7) | 97.6 (16.6)

7. Secondary Outcome: Low Density Lipoprotein Cholesterol (mg/dL)
Description: Measured in serum
Time Frame: Baseline, 4-weeks, 8-weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dietitian-Directed Diet Then Self-Directed Diet | Self-Directed Diet Then Dietitian-Directed Diet
Number analyzed (Participants) | 22 | 21
mg/dL
  Baseline | 109.0 (31.1) | 115.5 (41.2)
  Period 1 | 105.3 (34.4) | 113.4 (41.5)
  Period 2 | 107.5 (33.8) | 105.5 (36.8)

8. Secondary Outcome: Body Mass Index (kg/m^2)
Description: Derived from baseline height, and serial weight measurements
Time Frame: Baseline, 4-weeks, 8-weeks
Population: One person in the Dietitian-Directed Diet and then Self-Directed Diet did not provide a body mass index measurement during the follow-up visit.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Dietitian-Directed Diet Then Self-Directed Diet | Self-Directed Diet Then Dietitian-Directed Diet
Number analyzed (Participants) | 22 | 21
kg/m^2
  Baseline | 33.4 (6.4) | 33.5 (7.5)
  Period 1: number analyzed (Participants) | 21 | 21
  Period 1 | 33.0 (6.4) | 33.6 (7.8)
  Period 2: number analyzed (Participants) | 21 | 21
  Period 2 | 33.6 (6.5) | 33.5 (8.0)

ADVERSE EVENTS:
Time Frame: This was a crossover design of 2 interventions. Each intervention lasted about 4 weeks. Adverse events in response to the intervention were assessed at the end of each intervention period during an in-person visit. Thus adverse event surveillance was performed at 4 weeks and 8 weeks for each participant in the study.
Arm/Group | Dietitian-Directed Diet | Self-Directed Diet
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

LIMITATIONS AND CAVEATS:
There may have been carryover effects from the interventions on the primary outcome (serum urate). We were not adequately powered to rule out carry over effects, using a period-by-intervention interaction term in our models.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT03569020/ICF_000.pdf
  • Study Protocol (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT03569020/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT03569020/SAP_002.pdf